CLINICAL TRIAL: NCT07125872
Title: Open Label, Phase 2 Study of CD19t-haNK and N-803 in Combination With Rituximab in Participants With Relapsed/ Refractory B-cell Non- Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ResQ215A-BCELL
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-05

CONDITIONS: Relapsed B-Cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label- Single Arm (Other): Study is open label: combination of SOC Chemo therapy and investigational products.
  Interventions: Biological: CD19 t-haNK- IV Administration

INTERVENTIONS:
Biological: CD19 t-haNK- IV Administration — N-803 Subcutaneous (SQ): N-803 is a novel IL-15 superagonist immunotherapy administered subcutaneously. It is designed to enhance the proliferation and activation of natural killer (NK) cells and CD8+ T cells without stimulating regulatory T cells. N-803 SQ differs from other cytokine therapies due to its improved pharmacokinetic profile, enhanced in vivo activity, and reduced toxicity.
  CD19-Directed Therapies: CD19-targeted therapies, are biologic agents specifically designed to recognize and eliminate CD19-expressing B-cell malignancies. These therapies differ from traditional chemotherapy or small molecule inhibitors by leveraging the patient's immune system to achieve targeted cytotoxicity. Their mechanism of action involves direct binding to the CD19 antigen on malignant B cells, leading to immune-mediated cell death.

SUMMARY:
Open Label, Phase 2 Study of CD19t-haNK and N-803 in Combination with Rituximab in subjects with Relapsed/ Refractory B-cell Non- Hodgkin Lymphoma. 40 Participant will be screened for 20 subjects enrollment.

DETAILED DESCRIPTION:
Participants will receive treatment for a maximum of 12 cycles( 36 weeks) or until they have PD, unacceptable toxicity, withdrawal consent, or if the investigator feels it is no longer their best interest to continue treatment.

Subjects first receive chemo depletion chemo( Fludarabine and cyclophosphamide) for 3 consensual days, then subjects receive CD19t-haNK, N-803 and Rituximab every 3 weeks for up to 6 cycles. If subjects respond to treatment they will receive maintenance therapy from cycle 7 to 12. All participants should be followed for collection of survival statis, disease status, and posttreatment therapies every 12 weeks(+/- 2 weeks). The follow up visits may occur in-person or via phone contact.

Each cycle has day 1 and 8 for treatment. On day one of each cycle the following will be conducted: Concomitant Medication, Physical Exam, Vitals, ECOG and Labs. The participants will receive phone call 6 hours(+/-2) and 24 (+/-4 hours) and 24 post infusion for AE collection during cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age>18 years old 2- Able to understand and provide a signed informed consent that fulfills the relevant Human Research Ethics Committee( HRECC) or independent Ethics Committee( IEC) guidelines 3. Histologically or flow cytometry documented B-cell NHL, (excluding primary central nervous system [CNS] lymphoma, chronic lymphocytic leukemia [CLL], and Burkitt lymphoma) with the following specific criteria:

  * Have completed ≥2 lines of cytotoxic chemotherapy.
  * Have received rituximab or another anti-CD20 antibody.
  * Have measurable disease by Lugano classification documented within 8 weeks of the time of consent, defined as nodal lesions >15 mm in the long axis or extranodal lesions >10 mm in long and short axis, or bone marrow involvement that is biopsy proven.

    4. Eastern Cooperative Oncology Group (ECOG) performance status (Appendix 5) of 0 to 1.

    5. Stated willingness to comply with study procedures. 6. Able to attend required study visits and return for adequate follow-up, as required by this protocol.

    7. Agreement to practice effective contraception for female participants of childbearing potential and nonsterile males. Female participants of childbearing potential must agree to use effective contraception while on study and for at least 30 days after the last dose of study drug. Nonsterile male participants must agree to use a condom while on study and for up to 30 days after the last dose of study drug. Effective contraception includes orals, injectables, surgical sterilization (e.g., vasectomy, tubal ligation), two forms of barrier methods (e.g., condom, diaphragm) and implants such as intrauterine devices (IUDs).

Exclusion Criteria:

* Participants with ANY of the following criteria are excluded from participation in the study:

  1. Histologically documented primary CNS lymphoma, CLL, Burkitt, Burkitt-like lymphoma.
  2. Known hypersensitivity or allergy to any component of the study medications, including sulfa-containing study medication(s) (e.g., albumin [human], dimethyl sulfoxide [DMSO]).
  3. Inadequate organ function, evidenced by the following laboratory results:

     1. ANC < 1000 cells/mm3.
     2. Platelet count < 100,000 cells/mm3.
     3. Total bilirubin ≥ 1.5 × the upper limit of normal (ULN; unless the participant has documented Gilbert's syndrome or indirect hyperbilirubinemia).
     4. Aspartate aminotransferase (AST [SGOT])/ALT (SGPT) ≥ 2.5 × ULN.
     5. Alkaline phosphatase (ALP) levels ≥ 2.5 × ULN (or ≥ 5 × ULN in participants with bone metastases).
     6. Serum creatinine ≥ 160 µmol/L. NOTE: Each study site should use its institutional ULN to determine eligibility.
  4. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the participant at high risk for treatment-related complications.
  5. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon: such as systemic lupus erythematous, Wegner's glomerulonephritis, autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura requiring steroid therapy defined as > 20 mg of prednisone or equivalent daily.
  6. History of allogeneic hematopoietic stem-cell transplantation (HSCT) requiring ongoing systemic graft versus host disease (GvHD) therapy.
  7. Anti-CD20 antibody treatment less than 2 weeks prior to cell infusion.
  8. History of receiving allograft organ transplant requiring immunosuppression.
  9. Participants post solid organ transplants who develop high grade lymphomas or leukemias.
  10. Metastases to the CNS, including parenchyma or leptomeninges.
  11. Nonmalignant CNS disease (e.g., stroke, epilepsy, vasculitis, or neurodegenerative disease).
  12. History of active inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
  13. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (i.e., active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association (Appendix 6) Class 2 or higher; or serious cardiac arrhythmia requiring medication.
  14. Current chronic daily treatment (continuous for >3 months) with systemiccorticosteroids as defined as >20 mg of prednisone or equivalent daily, excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in participants who have known contrast allergies is allowed.
  15. Currently taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
  16. Tested positive for tuberculosis (TB) utilizing the QuantiFERON Gold TB test.
  17. History of human immunodeficiency virus (HIV) with current CD4+ T-cell count < 350 cells/μL and a detectable HIV viral load.
  18. Known carriers of hepatitis B virus (HBV) infection that is currently hepatitis B surface antigen (HBsAg) positive.
  19. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin.
  20. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
  21. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-19 (Estimated); Primary Completion 2027-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints( Efficacy) | 6 months
  ORR in accordance with Lymphoma Response to Immunomodulatory Therapy Criteria(LYRIC).
  OS( Time from study treatment initiation to death)

SECONDARY OUTCOMES:
Secondary endpoints( Safety) | 2 years
  Incidence of treatment- emergent adverse events( TEAEs) and serious adverse event(SAEs) graded using the National Cancer Institute( NCI) CTCAE Version 5.0, Clinically important changes in laboratory. Clinically important changes in vital sign Clinically important changes in laboratory tests Clinically important changes in vital signs

IPD SHARING:
Plan to Share IPD: Undecided